CLINICAL TRIAL: NCT00993811
Title: The Shang Ring: A Novel Male Circumcision Device for HIV Prevention
Acronym: ShangRing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: EngenderHealth (Other)
Responsible Party: Marc Goldstein, M.D., Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0902010241
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2009-10

CONDITIONS: Male Circumcision; HIV Prevention; HIV Infections
Keywords: male circumcision; HIV; Africa; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Circumcision (Experimental): Males undergoing circumcision
  Interventions: Device: Shang Ring circumcision

INTERVENTIONS:
Device: Shang Ring circumcision — novel device for adult male circumcision
  Other Names: adult male circumcision

SUMMARY:
The purpose of this study is to evaluate the Shang Ring, a novel Chinese device for voluntary medical male circumcision, in order to improve the provision of male circumcision services for HIV prevention in Africa.

DETAILED DESCRIPTION:
Three randomized clinical trials (RCTs) have confirmed the benefit of voluntary medical male circumcision (VMMC) in reducing the acquisition of HIV by circumcised men. In Africa, VMMC is most commonly performed with the methods described in the WHO Manual for Male Circumcision under Local Anaesthesia (i.e., the forceps-guided, dorsal slit or sleeve method).

Modelers have estimated that to scale-up VMMC to prevent large numbers of HIV infections will require millions of circumcisions over the next 5 to 10 years, with more than 10 million circumcisions in 2012 based on aggressive scale-up plans.

Neonatal circumcision is a very common procedure and has been the subject of numerous clinical trials. With the use of simple devices, neonatal circumcision is rapid and safe. In contrast, current adult surgical techniques are done freehand. Adolescent or adult male medical circumcision has been a rarely performed procedure in most developed countries. Circumcision has suffered from little or no research that could make possible either (a) comparison or simplification of surgical techniques or (b) development of devices to facilitate the procedure. Current techniques are time consuming and require long training periods to produce skilled personnel. Each procedure typically takes 20 to 40 minutes.

A search for more efficient adult circumcision techniques has been undertaken by consultants for the World Health Organization (WHO) and the Bill & Melinda Gates Foundation. Preliminary discussions that helped to produce this proposal suggest that the Shang Ring is one of the most promising existing devices that could greatly simplify adult circumcision. More efficient and simpler techniques could potentially:

* Reduce the operating time and the cost of supplies
* Improve the safety of the procedure
* Permit more rapid training of non-physician health care providers
* Accelerate the process of scaling up this proven HIV prevention strategy

The Shang Ring is a relatively new device, manufactured by SNNDA, a small company based in Wuhu, China owned by Mr. Shang Jianzhong Shang. It has been approved for marketing in China since 2005, with sales of about 40,000 devices in the past couple of years. The Shang Ring and was awarded the CE Mark by for the European Union in October, 2008. The Shang Ring has the potential to dramatically reduce the time needed for the surgical procedure, from the current 20 to 430 minutes, to an average of about 5 3 to 10 minutes per procedure. This efficiency would greatly increase the productivity of large scale VMMC efforts.

The Shang Ring has several unique advantages compared to other devices that are currently in use, including its suitability for use in adults, small size, simple design, and ease of application. It is a clamp- type device, so there is no need for cautery for hemostasis,, or for suturing for hemostasis, or wound closure. The manufacturer has agreed to negotiate a low public sector price so that it would be affordable for circumcision programs in Africa.

Project goal, objectives and critical milestones: We propose to conduct a multicenter RCT comparing the Shang Ring to standard surgical techniques, with a sample size of 500 men in the Shang Ring group and 500 men in the standard surgery group. We will conduct cost studies to compare time and resources needed for both techniques. We will also assist SNNDA in preparing and submitting dossiers to regulatory authorities in both the United States and at least three African countries, and will assist as needed in SNNDA's application to the U.S. FDA for 510(k) clearance. Circumcision devices are considered class II devices by the U.S. FDA. We will request that the FDA grant marketing clearance for the Shang Ring through a 510(k) process, similar to other recent circumcision device approvals. We propose to conduct these activities over a 30-month period. If successful, they could lead to wide use of the Shang Ring and dramatic efficiencies in scaling up VMMC programs.

ELIGIBILITY:
Inclusion Criteria:

* Freely consents to participate in the study and signs an informed consent form
* Ages 18 - 54 years
* Uncircumcised
* Good general health
* HIV sero-negative
* Able to understand the study procedures and requirements
* Agrees to return to the health care facility for the full schedule of follow-up visits after his circumcision

Exclusion Criteria:

* Previous circumcision on examination
* Age < 18 years or > 54 years
* Active genital infection, anatomic abnormality or other condition, which in the opinion of the surgeon prevents the man from undergoing a circumcision
* HIV sero-positive
* A condition, which in the opinion of the surgeon contradicts participation in the study

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The efficacy and safety of the ShangRIng device for adult male circumcision in an HIV endemic region in Africa. | Six week post-operative follow up appointment and examination

SECONDARY OUTCOMES:
Behavior outcomes (surgical acceptability, satisfaction, problems encountered with the device, compliance with post-surgical instructions, and correct knowledge about the extent of the protective effect of circumcision and safe sex). | Six week post-operative follow up appointment and examination

CONTACTS AND LOCATIONS:
Overall Officials: Mark Barone, DMD, Study Director — EngenderHealth; Marc Goldstein, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Homa Bay District Hospital, Homa Bay, Kenya